CLINICAL TRIAL: NCT06447467
Title: Short Term Outcome of Acute Heart Failure in Diabetic and Non Diabetic Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mena Monir Thabet, Resident at Internal medicine departement Sohag Universirty Hospital, Sohag University
Other Study IDs: Soh-Med-24-05-13MS
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Acute Heart Failure; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic patients: Diabetic patients
  Interventions: Diagnostic Test: pro BNP
- Non Diabetic patients: Non Diabetic patients
  Interventions: Diagnostic Test: pro BNP

INTERVENTIONS:
Diagnostic Test: pro BNP — Test is mainly used to help diagnose or rule out heart failure in a person who is having symptoms

SUMMARY:
Around 26 million people suffer from heart failure (HF) globally, and the prevalence is increasing with an increasing longevity, prevalence of risk factors, and improved survival in patients with cardiovascular diseases In Egypt, HF is the primary cause of hospitalization among patients aged > 65 years . Hospitalization for HF is associated with a high mortality and rate of re-hospitalization . Around 75% patients with HF have ≥ 1 comorbidity, and these comorbidities make overall clinical outcomes worse . In a recent meta-analysis, patients with diabetes mellitus (DM) were suggested to have a two-fold increase in the risk of HF . DM is present in ~ 35% patients hospitalized with acute HF . Multiple factors such as ischemia, hypertension, and extracellular fluid volume expansion are involved in the pathogenesis of HF in DM.

DETAILED DESCRIPTION:
The prevalence of both heart failure (HF) and diabetes has increased over the last decades and is expected to do so in the upcoming decades . Therefore, the presence of diabetes in patients with HF is also likely to increase and this is anticipated to become a major health concern. The actual prevalence of diabetes in patients with acute HF in different registries has varied but may be as high as 45% . Because the structure and function of the heart is directly influenced by the presence of diabetes, diabetes is to be considered to represent more than just a co morbid condition in HF .

Diabetes has been shown to be an independent risk factor for the development of HF . Moreover, this risk has been shown to be age and sex dependent. Compared with patients without diabetes, the presence of diabetes doubles the risk of HF in men, and the risk of developing HF in women may be as much as four times higher . These associations may even be stronger in younger patients. Furthermore, the presence of diabetes has been associated with a longer duration of hospitalization and higher rates of rehospitalization among patients with acute HF. Importantly, in patients with HF, it has been established that the presence of diabetes is not only associated with an increased cardiovascular morbidity but also with an increased mortality

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or older .
* Admitted to the Coronary Care Unit with acute HF.
* Patients with new onset heart failure.
* Decompensated chronic HF.

Exclusion Criteria:

* Aged under 18 years old.
* Patients with chronic HF

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Aged 18 years old or older .
  * Admitted to the Coronary Care Unit with acute HF.
  * Patients with new onset heart failure.
  * Decompensated chronic HF.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pro BNP level | 6 months
  A pro BNP test is mainly used to help diagnose or rule out heart failure in a person who is having symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Magdy M Amin, Professor, Principal Investigator — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bui AL, Horwich TB, Fonarow GC. Epidemiology and risk profile of heart failure. Nat Rev Cardiol. 2011 Jan;8(1):30-41. doi: 10.1038/nrcardio.2010.165. Epub 2010 Nov 9. PMID 21060326
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Ambrosy AP, Fonarow GC, Butler J, Chioncel O, Greene SJ, Vaduganathan M, Nodari S, Lam CSP, Sato N, Shah AN, Gheorghiade M. The global health and economic burden of hospitalizations for heart failure: lessons learned from hospitalized heart failure registries. J Am Coll Cardiol. 2014 Apr 1;63(12):1123-1133. doi: 10.1016/j.jacc.2013.11.053. Epub 2014 Feb 5. PMID 24491689
- [Background] Cook SA, Varela-Carver A, Mongillo M, Kleinert C, Khan MT, Leccisotti L, Strickland N, Matsui T, Das S, Rosenzweig A, Punjabi P, Camici PG. Abnormal myocardial insulin signalling in type 2 diabetes and left-ventricular dysfunction. Eur Heart J. 2010 Jan;31(1):100-11. doi: 10.1093/eurheartj/ehp396. Epub 2009 Oct 1. PMID 19797329